CLINICAL TRIAL: NCT00815464
Title: Efficacy Study of Liquid Acupuncture(Herb Acupoint Injection) Therapeutics in Chronic Hepatitis B(CHB) Based on Patients' Individual Condition
Brief Title: A Single-Arm Study Evaluating the Efficacy of Liquid Acupuncture Therapeutics in Chronic Hepatitis B
Acronym: CHB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yu Medical Garden (Other)
Responsible Party: Yu, Ke Heng / Registered Medical Practitioner, Yu Medical Garden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMG-PR-001
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Hepatitis B, Chronic; Liver Diseases; Virus Diseases; Hepatitis; Diffuse Hepatic Disease
Keywords: Chronic Hepatitis B; Liquid Acupuncture(Herb Acupoint Injection); Therapeutics; Herbalist; Acupoint
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Diseases; Virus Diseases; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antiviral Therapy (Experimental): Liquid Acupuncture(Herb Acupoints Injection) Therapeutics was researched and developed by Herbalist Yu Ru Lin in early of 1950s and used by Yu Medical Garden till now. It is an integrated therapeutics,according to individual condition, select the Acupoints(not limit to current used common acupoints) and proper herbs made individually.It is a special medical treatment conception, which theory is utilizing patients' condition, mobilizing their individual internal curability,therefore the final efficacy can be retrieved.
  Interventions: Device: Liquid Acupuncture (Herb Acupoint Injection)

INTERVENTIONS:
Device: Liquid Acupuncture (Herb Acupoint Injection) — Each 4 weeks per one circle.The first 3 weeks for treatment practice(one per week)and the last week for test collection.
  Other Names: Antiviral Agents

SUMMARY:
Study Purpose:

The purpose of this study is to assess that Liquid Acupuncture(Herb Acupoints Injection) Therapeutics could achieve permanent efficacy response in Chronic Hepatitis B.

Efficacy Assessment:

At cessation of the Treatment(about at 24 weeks)comparing Testing Data with the Normal Criteria and their individual baseline.Continue for monitoring the Status 1-5 years.

Data Analysis:

Each 4 weeks collecting Patients' testing data and fill a table.A summary table will be presented as frequency tables for categorical variables as number or percentage.

DETAILED DESCRIPTION:
Inclusion Criteria & Outcome:

Documented chronic hepatitis B infection positive serum HBV-DNA 10^5 copies/mL & above.

Permanent efficacy response after whole treatment circle close(about 24 weeks,someone may be later than 24 weeks but within 48 weeks)

* HBeAg loss(if HBeAg positive)
* Liver Function normal(if Liver Function off normal)
* HBV DNA non-detectability (PCR <500 copies/ml)
* Image of chronic diffuse hepatic disease will recover up to normal if have.
* HBsAg titer will decrease continually up to loss after cessation of the treatment.

Treatment Procedure:

Patients will be involved in the study for up to 24-48 weeks from enrollment. There is no external sponsor, commercial sponsor nor governmental agency on this study. The study will be conducted only by Dr. Yu, Ke Heng,who is master of the Liquid Acupuncture(Herb Acupoint Injection)practice more than 30 years.About 30 subjects will be involved in the study overall. All the subjects can be filled up worldwide.

Patients will be required to rent apartment or house for staying at the city(Xiamen city,China preferred).Dr. Yu will go to the Patients' site for treatment practice weekly,each 4 weeks is one circle(the first 3 weeks for treatment practice and last week for Test collection).Appointed Hospitals for test must be certificated and qualified(Chang Gang Hospital preferred).Dr. Yu will explain the test results individually.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-55 years inclusive.
* Documented chronic hepatitis B infection determined by the presence of serum HBsAg for at least 6 months.
* Serum HBV DNA ≥ 10^4 copies/mL(PRC).
* Use of interferon alfa, thymosin, or antiviral agents less than 1 year and not receive them more than 2 months. (If you expect to stop these agents but worry about the risk, you may ask us to help.)
* Agree not to participate in any other investigational trials or to undertake other HBV systemic antiviral regimens during participation in this study.
* Able to give written informed consent and comply with the requirements of the study.

Exclusion Criteria:

* Superinfection/Coinfection with hepatitis A, hepatitis C, hepatitis D, hepatitis E or HIV.
* Autoimmune hepatitis (antinuclear antibody titre > 1:160).
* Use of interferon alfa, thymosin, or antiviral agents more than 1 year.
* Pregnant or nursing.
* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include, may not limit to, renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, active infection or cancer.
* Clinical signs of decompensated liver disease at baseline. These may include but are not limited to:serum bilirubin > 2.5 mg/dL (≤ 43 µmol/L), prothrombin time > 2 second prolonged above ULN,serum albumin < 35g/L,history of ascites, variceal bleeding, or encephalopathy,Alanine aminotransferase (ALT) >10 times ULN at screening or history of acute exacerbation leading to transient decompensation.
* Hepatocellular carcinoma as evidenced by one of the following:

  * suspicious foci on ultrasound or radiological examination.
  * where no positive ultrasound finding, but serum alpha-fetoprotein > 100ng/mL
  * Active alcohol or drug abuse or history of alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
* Received hepatotoxic drugs (e.g., anabolic steroids, ketaconazole, itraconazole, isoniazid, rifampin, rifabutin) within 2 months prior to study screening or expected to receive these during the course of the study.
* Received nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine etc.) or competitors of renal excretion (e.g., probenecid) within 2 months prior to study screening or the expectation that patient will receive any of these during the course of the study.
* Receiving systemic (intravenous or oral) steroids, immuno-suppressant therapies or chemotherapeutic agents within 2 months of study screening or expected to receive these agents during the course of the study.
* Neutrophile granulocyte count <1.0*10e9/L and Platelet count < 30*10e9/L.
* Inability to comply with study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Permanent Efficacy response after whole treatment circle close(about 24-48 weeks): 1、HBeAg loss(if HBeAg positive) 2、HBV DNA non-detectability (PCR <500 copies/ml) 3、Liver function normal(If Liver function off normal) | 1-2 years

SECONDARY OUTCOMES:
HBsAg titer will decrease continually up to loss after cessation of the treatment. | one year later

CONTACTS AND LOCATIONS:
Overall Officials: Ke Heng Yu, Principal Investigator — Yu Medical Garden